CLINICAL TRIAL: NCT02757469
Title: Drospirenone and Ethinyl Estradiol Combinations (Yasmin) as Infertility Treatments for Premature Ovarian Failure: a Perspective Follow-up Study.
Brief Title: Oral Contraceptives as Infertility Treatments for Premature Ovarian Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Yunhai Chuai, Department of Obstetrics and Gynecology, Navy General Hospital, Beijing, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCPOF-1
Record Dates: First submitted 2016-04-24; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Primary Ovarian Insufficiency; Menopause, Premature
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature | interventions — drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yasmin (Experimental): Pregnancies will occur while the women are taking oral contraceptives (Yasmin). The possible role of exogenous estrogens in sensitizing the granulosa cells to the effect of follicle-stimulating hormone and thereby inducing ovulation and conception in some women with premature ovarian failure is examined.
  Interventions: Drug: Drospirenone and ethinyl estradiol combination (Yasmin)

INTERVENTIONS:
Drug: Drospirenone and ethinyl estradiol combination (Yasmin) — Female oral combined contraceptive containing 30 mcg (0.030 mg) Ethinyl Estradiol and 3 mg drospirenone (Androstenes)

SUMMARY:
Premature ovarian insufficiency (POI) is a life-changing condition that affects women in their reproductive age. There is a lack of reports which focus on how to improve the reproductive outcome of these women who wish to conceive spontaneously or use assisted conception with their own oocytes. However, one could surmise that it is important to lower gonadotropin levels into the physiological range before embarking on any treatment, even if natural conception is the only choice for the woman/couple.

ELIGIBILITY:
Inclusion Criteria:

* premature ovarian failure
* normal anatomy
* normal secondary sexual characteristics
* essential or idiopathic

Exclusion Criteria:

* chromosomal disorder
* iatrogenic injury
* autoimmune diseases
* infection
* genetic diseases

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
live birth | 3 years
  The event that a FETUS is born alive with heartbeats or RESPIRATION regardless of GESTATIONAL AGE. Such liveborn is called a newborn infant (INFANT, NEWBORN).

SECONDARY OUTCOMES:
clinical pregnancy rate | 3 years
  The ratio of the number of conceptions (CONCEPTION) including LIVE BIRTH; STILLBIRTH; and fetal losses, to the mean number of females of reproductive age in a population during a set time period.
multiple pregnancy | 3 years
  The condition of carrying two or more FETUSES.
miscarriage | 3 years
  Expulsion of the product of FERTILIZATION before completing the term of GESTATION and without deliberate interference.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shang, Dr, Principal Investigator — Navy General Hospital, Beijing
Locations (1):
- Navy General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Alper MM, Jolly EE, Garner PR. Pregnancies after premature ovarian failure. Obstet Gynecol. 1986 Mar;67(3 Suppl):59S-62S. doi: 10.1097/00006250-198603001-00018. PMID 3080719
- [Result] Ben-Nagi J, Panay N. Premature ovarian insufficiency: how to improve reproductive outcome? Climacteric. 2014 Jun;17(3):242-6. doi: 10.3109/13697137.2013.860115. Epub 2013 Dec 16. PMID 24341612